CLINICAL TRIAL: NCT01042067
Title: Safer Warfarin Treatment - the Influence of CYP2C9 Genotyping, Genotyping of Vitamine K Dependent Proteins and Dietary Vitamine K Status on Dosing, Clinical Effect and Adverse Events With Emphasis on the Initial Phase of Treatment
Brief Title: Safer Warfarin Treatment
Acronym: CYKOWAR
Status: Suspended | Type: Observational
Why Stopped: Enrolling participants has halted due to lack of investigator.
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Norwegian Medicines Agency (Other Government); Norway: South-Eastern Norway Regional Health Authority (Unknown)
Other Study IDs: 2006-001895-18
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Atrial Fibrillation; Venous Thrombosis; Pulmonary Embolism; Heart Valve Prosthesis
Keywords: warfarin; genotyping; vitamin K; dosing; adverse events; initial phase of treatment; algorithm
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Warfarin treatment group: Open label study. Patients in need of warfarin treatment (standard indications) are included in the study at the onset of warfarin treatment.
  Interventions: Other: Blood specimens (whole blood, serum, plasma)

INTERVENTIONS:
Other: Blood specimens (whole blood, serum, plasma) — The patients follow standard warfarin treatment regimens and the only intervention is the sampling of blood specimens.

SUMMARY:
The study is a national multicenter prospective observational study, including 200 patients. The main purpose of this study is to explore in more detail the influence of genetic variability (CYP enzymes and vitamin K dependent proteins) and dietary vitamin K status on warfarin dosing, clinical effect and adverse events with emphasis on the initial phase of treatment. The hypothesis is that genetic variability concerning CYP enzymes and vitamin K dependent proteins predict dosing and adverse events during warfarin treatment. The main aim is to individualize warfarin therapy and establish a treatment algorithm based on genotype and dietary vitamin K status to make the anticoagulation therapy with warfarin more secure.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* >18 years of age
* included in the study at the onset of warfarin treatment
* target INR (2-3 for atrial fibrillation, vein thrombosis, pulmonary embolism and 2.5-3.5 for prosthetic heart valves)
* standard indications for warfarin treatment

Exclusion Criteria:

* Non-caucasian
* Clinical significant liver affection
* Heart failure, NYHA class III-IV
* Non-compliant - not able to accomplish protocol demands
* Not able to give informed consent
* Long-term antibiotic therapy
* Malabsorption conditions and inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of warfarin treatment (standard indications) are included in the study at the onset of warfarin treatment. About 200 patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-01

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway